CLINICAL TRIAL: NCT03321825
Title: Evaluation of the Merz Cheek Fullness Assessment Scale in the Treatment of Midface Volume Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930071002
Record Dates: First submitted 2017-10-04; First posted 2017-10-26 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Moderate to Severe Midface Volume Deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belotero® Volume Lidocaine (Experimental): Subdermal injection
  Interventions: Device: Belotero® Volume Lidocaine
- No treatment (No Intervention)

INTERVENTIONS:
Device: Belotero® Volume Lidocaine — Mode of application: subdermal injection
  Other Names: Hyaluronic acid dermal filler containing 0.3% of lidocaine hydrochlorid
  Arms: Belotero® Volume Lidocaine

SUMMARY:
Evaluation of the sensitivity of the Merz Cheeks Fullness Assessment Scale (MCFAS) and the clinical relevance of aesthetically pleasing outcomes by detecting changes in cheek appearance after Belotero® Volume Lidocaine injection.

The safety objectives include the identification and description of adverse events (AEs), adverse device effects (ADEs), serious adverse events (SAEs), serious adverse device effects (SADEs), anticipated serious adverse device effects (ASADEs) and unanticipated adverse device effects (UADEs) during the course of the study. Additionally, common treatment site responses (CTRs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has right and left cheek volume deficit with a rating of 2 or 3 (moderately or severely sunken cheeks) on the MCFAS as determined by the blinded evaluator.
* 2. Has the same MCFAS score on both cheeks (i.e., cheeks are symmetrical).
* 3. Is at least 18 years of age.
* 4. Understands and accepts the obligation not to receive any other procedures (i.e., dermal fillers, toxin treatments, facial ablative or fractional laser, microderm abrasion, chemical peels, non-invasive skin-tightening [e.g., Ultherapy, Thermage] and/or surgical procedures) in the face during participation in the study.

Exclusion Criteria:

* 1. Skin atrophy in the midfacial region other than that related to age.
* 2. Has gained or lost and ≥ 2 body mass index (BMI) units within the previous 90 days or has the intention to gain or lose a significant amount of weight during the course of the study.
* 3. Unphysiological skin laxity and/or sun damage beyond typical for the subject's age or subject plans to tan during the study period.
* 4. Acute inflammatory process or infection at the injection site (e.g., acne, eczema, streptococcus infections), or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of AEs.
* 5. Prior surgery, including midfacial plastic surgery, or has a permanent implant or graft in the midfacial region that could interfere with effectiveness assessments.
* 6. Undergone oral surgery in the past 30 days or plans to undergo oral surgery during participation in the study (i.e., orthodontia, extraction, implants).
* 7. Ever been treated with fat injections or permanent and/or semi-permanent dermal fillers in the midfacial region or plans to receive such treatments during participation in the study.
* 8. Received midfacial region treatments with porcine-based collagen fillers or with Belotero Volume, JUVÉDERM VOLUMA®, or Restylane® Lyft, calcium hydroxylapatite (CaHA), poly L-lactic acid (PLLA), or mesotherapy within the past 24 months and/or with other hyaluronic acid (HA) products within the past 12 months or plans to receive such treatments during participation in the study.
* 9. Received facial dermal therapies (i.e., toxin treatments, facial ablative or fractional laser, microderm abrasion, chemical peels, non-invasive skin-tightening [e.g., Ultherapy, Thermage] and surgical procedures) in the midface region within the past 12 months or plans to receive them during participation in the study.
* 10. Facial nerve palsy or history of facial nerve palsy.
* 11. A history or documented evidence of an autoimmune disease (e.g., scleroderma, lupus erythematosus, rheumatoid arthritis).
* 12. A known bleeding disorder or has received or is planning to receive anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs (e.g., aspirin, ibuprofen), or other substances known to increase coagulation time (vitamins or herbal supplements, e.g., vitamin E, garlic, gingko), from 10 days before to 3 days after injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the responder rate between the treatment group and the untreated control group at Week 4, according to the Merz Cheeks Fullness Assessment Scale (MCFAS) as assessed by a blinded evaluator. | Week 4
  Treatment response is defined as ≥ 1-point improvement on both cheeks compared to baseline.
  The MCFAS is a 5-point ordinal rating scale ranging from 0 (full cheek) to 5 (very severely sunken cheek).

SECONDARY OUTCOMES:
Descriptive summary of the FACE-Q satisfaction of the midface for treated subjects at baseline and Week 4 | Week 4
  Subject's assessment is based on the entire face. FACE-Q scores are derived from questionaires 'satisfaction with cheeks' (including 5 questions relating to the satisfaction with cheek appearance, answers range from 1 (very dissatisfied) to 4 (very satisfied)), and the module 'patient-perceived age visual analogue scale' (VAS - scale ranging from -15 (15 years younger) to 15 (15 years older)).
Average percent change of the FACE-Q satisfaction of the midface for treated subjects from baseline to Week 4 | Week 4
  Subject's assessment is based on the entire face. FACE-Q scores are derived from questionaires 'satisfaction with cheeks' (including 5 questions relating to the satisfaction with cheek appearance, answers range from 1 (very dissatisfied) to 4 (very satisfied)), and the module 'patient-perceived age visual analogue scale' (VAS - scale ranging from -15 (15 years younger) to 15 (15 years older)).
Descriptive summary of Global Aesthetic Improvement Scale (GAIS) scores for treated subjects at Week 4, as completed by the treating investigator. | Week 4
  This assessment is a measure of aesthetic improvement relative to the baseline, pre-treatment condition, as assessed from photographs.
  The Investigator-GAIS is a 7-point scale ranging from -3 (very much worse) to +3 (very much improved).
Descriptive summary of GAIS scores for treated subjects at Week 4, as completed by the subject. | Week 4
  This assessment is a measure of aesthetic improvement relative to the baseline, pre-treatment condition, as assessed from photographs.
  The Investigator-GAIS is a 7-point scale ranging from -3 (very much worse) to +3 (very much improved).
Evaluate the incidence and nature of device- and/or injection-related AEs, and SAEs observed during the study. | Week 4
Common treatment site responses (CTRs) will be evaluated using subject diaries | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Merz Scientific Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (3):
- Canada (3):
  - Institute of Cosmetic and Laser Surgery; Merz Inverstigational Site #0010409, Oakville, Ontario
  - Research Toronto; Merz Investigational Site #0010408, Toronto, Ontario
  - Cosmetic Dermatology Toronto Yorkville; Merz Investigational Site #'0010412, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No